CLINICAL TRIAL: NCT02603211
Title: Tactile Breast Imaging Sensor for Tumor Malignancy Characterization
Status: Completed | Type: Observational
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Other Study IDs: 22050
Record Dates: First submitted 2015-11-03; First posted 2015-11-11 (Estimated); Results first posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with Breast Tumors: Women with breast tumors.
  Interventions: Device: tactile imaging sensor or system made in our laboratory

INTERVENTIONS:
Device: tactile imaging sensor or system made in our laboratory — This is a camera with elastomer tip and LED lights. It is a harmless device.
  Other Names: mechanical property estimation device; tactile sensor

SUMMARY:
The aim of this study is to see how well a tactile imaging sensor will detect for breast masses compared to traditional mammography and/or ultrasound. This device may allow a simple, convenient method to screen for breast tumors. This data will be used to check the feasibility of using the device to detect breast tumors.

DETAILED DESCRIPTION:
The tactile imaging sensor will estimate the relative size and elasticity of the mass(es). This device may allow a simple, convenient method to screen for breast tumors. This is not a treatment and it will not be used to diagnose abnormal masses. The investigators will also not look for any unknown masses. And only doctors will touch the patients. An engineering assistant will be in the room to operate the tactile imaging sensor.

The breast scan that is done as part of this research protocol is not intended to detect any breast disease or abnormality. Research breast scans are not examined by a clinical radiologist to look for abnormalities. Research scan will be evaluated by the engineers developing the device to assess its usefulness. The breast scan for this research will only look at a portion of your breast as it relates to this research. The investigators, the tactile imaging sensor operators and other members of the research team are not qualified to interpret the scan for any diagnostic or therapeutic value. Therefore, the tactile imaging scan being done for this research study will not be analyzed to detect any medical condition.

Patients will have done mammography or ultrasound by now. Once the doctor decides to perform biopsy, the tactile imaging will be planned. The consent will be obtained before the biopsy. One of the investigators (Dr. Caroline or Dr. Reilly) will obtain the consent. Before the biopsy, the doctor will identify the mass(es) using other modalities such as a ultrasound. The tactile imaging sensor operator will obtain the tactile images. Then the biopsy will be performed. Radiology doctor, resident, and radiology technologist are always present during the procedure. In addition a professional assistant from the engineering group will operate the tactile imaging sensor. That person will not have any physical contact with you. The procedure will be very similar to the ultrasound device.

The images will be analyzed by the investigators.

ELIGIBILITY:
Inclusion Criteria:

* Women who had mammogram and/or ultrasound birads (category IV or V)
* Women ages between 30 and 80.
* Women who have been scheduled for biopsy from the Temple breast surgery clinic
* Women who have been scheduled for biopsy by Dr. Kathleen Reilly.
* Women, who speak and understand English.

Exclusion Criteria:

* Women who do not meet the criteria requiring biopsy.
* Women who have allergic reaction to silicone.
* Women who cannot speak or understand English.
* Women who are pregnant.
* Women, younger than 30 years old, and older than 80 years old.

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who had mammogram and are getting biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-03-11 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2017-10-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Women With Breast Tumors
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Women With Breast Tumors
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Size Error in Millimeters
Description: We obtain the image of the tumor and estimate its size. We compare this with the mammogram size data to compute the size error.
Time Frame: 1 year
Measure: Mean (Standard Error); unit: milimeters
Groups:
- Women With Breast Tumors: Women with breast tumors, who come for biopsy are recruited for this study.
Arm/Group | Women With Breast Tumors
Number analyzed (Participants) | 20
milimeters | 0 (5)

2. Secondary Outcome: Malignancy Estimation Using Risk Score
Description: The tumor risk score is calculated from the tumor size and deformation index. The scale will be from 0 to 5. With 0 being likely to be benign and 5 being likely to be malignant.
  We weigh the size 30% and deformation index 70% to come with the risk score. The tumor size is given in millimeters and deformation index is unitless.
  Deformation Index represents the hardness of the tumor. The amount at which the probe tip gets deformed by applying a force is called deformation index.
  Under the condition that the applied force, depth of the tumor and size of the tumor phantom are kept constant, the softer tumor makes the probe tip deform less than the stiffer tumor. Hence the deformation index for stiffer inclusion will be higher than the softer tumors.
Time Frame: 1 year
Measure: Number; unit: participants
Groups:
- Women With Breast Tumors: Women with breast tumors who come for biopsy are recruited.
Arm/Group | Women With Breast Tumors
Number analyzed (Participants) | 20
participants | 2.0
Statistical Analysis 1: Comparison: Women With Breast Tumors; Test type: Other; We will obtain 20 tactile image data sets from the breast tumor patients. The tactile images will be converted to size and deformation index. Then these two parameters will be converted to the risk score. This is a small number of patients for statistically significance study. Therefore, we plan to use the Leave-One-Out-Cross-Validation (LOOCV) technique to validate the human test results to determine the performance of the device. We obtain the Risk Score. Risk Score is a unit less numerical value, which can be used as a scale to classify the tumor as malignant and benign. Based on the calculated size of the tumor and measured deformation index, the breast tumors are classified as benign and malignant using scoring method. The risk score will range from 0 to 5, where 0 represents the benign and 5 represents the malignant tumor. Comparing the Risk Score and the Pathology reports we obtain sensitivity, specificity and accuracy of the system

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Women With Breast Tumors
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT02603211/Prot_SAP_000.pdf